CLINICAL TRIAL: NCT04421586
Title: VISTA: Vaccinator-Initiated Screening and TAilored Counseling for Reducing Vaccine Hesitancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00100032
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-03

CONDITIONS: Vaccination Uptake
Keywords: vaccine hesitancy
MeSH Terms: conditions — Vaccination Hesitancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregnant women receiving VISTA counseling (Experimental): Up to 30 pregnant women are screened and counseled for vaccine concerns using VISTA
  Interventions: Behavioral: VISTA
- Pregnant women receiving usual care (No Intervention): Up to 30 pregnant women receiving usual care

INTERVENTIONS:
Behavioral: VISTA — VISTA will be an educational intervention.
  Arms: Pregnant women receiving VISTA counseling

SUMMARY:
The purpose of this study is to understand why parents do or do not vaccinate their children and explore what information parents need to vaccinate their children. The study will test whether information about vaccinations provided during pregnancy by a health provider (VISTA intervention) may improve the possibility that a child is vaccinated on time.

DETAILED DESCRIPTION:
The study will be implemented in 10 health facility catchment areas in Mtwara region, Tanzania. The study sites will be non-randomly assigned to receive VISTA or usual care.

Only core messages were developed and evaluated in this study. Tailored messages will be developed and evaluated in a follow-up study.

ELIGIBILITY:
Inclusion Criteria:

Study outcomes will be measured for health providers implementing the intervention and pregnant women receiving the intervention. Up to 10 health workers (including community health workers (CHW) from each of the intervention sites will participate in the study.

To participate in the study,

Health workers must be:

* 18 years of age or older
* Work in one of the study intervention sites

Women must be:

* In the third trimester of pregnancy
* Residing in a study site (intervention or control)
* At least 15 years of age
* Planning to reside in the study site for the duration of their participation in the study (until approximately 6 months after delivery to enable follow up).
* Have at least 1 concern about childhood vaccines

Exclusion Criteria:

There are no exclusion criteria.

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lavanya Vasudevan, PhD, Principal Investigator — Duke University
Locations (1):
- National Institute for Medical Research (NIMR), Mtwara, Tanzania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from medical clinics and surrounding communities in rural areas.
Units Other Than Participants: study sites
Groups:
- Pregnant Women Receiving VISTA Counseling: Up to 30 pregnant women are screened and counseled for vaccine concerns using VISTA (Vaccinator-Initiated Screening and TAilored Counseling for Reducing Vaccine Hesitancy)
  VISTA: VISTA will be an educational intervention.
Period: Overall Study
Arm/Group | Pregnant Women Receiving VISTA Counseling | Pregnant Women Receiving Usual Care
Started | 30; 5 study sites | 30; 5 study sites
Completed | 25; 5 study sites | 24; 5 study sites
Not Completed | 5; 0 study sites | 6; 0 study sites
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 2 | 2
Not completed — Withdrawn by PI | 1 | 0
Not completed — Infant death (no follow up data or vaccination outcomes) | 2 | 3

BASELINE CHARACTERISTICS:
Population: Participants on whom baseline/demographic data was collected.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregnant Women Receiving VISTA Counseling | Pregnant Women Receiving Usual Care | Total
Number analyzed (Participants) | 29 | 30 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.28 (7.04) | 28.10 (8.38) | 29.66 (7.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 30 | 59
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 29 | 30 | 59
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 30 | 59
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Tanzania | 29 | 30 | 59

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Women With Reduced Number of Concerns Immediately Post-counseling in the Intervention Arm
Time Frame: Post-counseling (Baseline visit)
Population: Outcome measure only applies to the VISTA arm.
Measure: Number; unit: percentage of women
Arm/Group | Pregnant Women Receiving VISTA Counseling | Pregnant Women Receiving Usual Care
Number analyzed (Participants) | 29 | 0
percentage of women | 51.72 |

2. Secondary Outcome: Percentage of Women With Reduced Number of Concerns in Intervention Versus Control Arms at Follow up.
Time Frame: Follow-up (up to 6 months post-birth; up to 9 months post-baseline)
Population: Data not collected on 6 participants in each group.
Measure: Number; unit: percentage of women
Arm/Group | Pregnant Women Receiving VISTA Counseling | Pregnant Women Receiving Usual Care
Number analyzed (Participants) | 25 | 24
percentage of women | 48.0 | 62.5

3. Secondary Outcome: Percentage of Children by Vaccine Who Received the Vaccine Within 4-week Window of Due Date in Intervention Versus Control Arm
Description: Includes early doses up to 1 week prior to due date. In the event of twins, information for only 1 child per mother was included in the determination of outcomes.
Time Frame: Follow-up (up to 6 months post-birth; up to 9 months post-baseline)
Population: Data not collected on 13 participants.
Measure: Number; unit: percentage of children
Arm/Group | Pregnant Women Receiving VISTA Counseling | Pregnant Women Receiving Usual Care
Number analyzed (Participants) | 25 | 23
percentage of children
  BCG | 96.00 | 86.96
  Polio 0 | 88.00 | 82.61
  Polio 1 | 64.00 | 73.91
  Polio 2 | 48.00 | 56.52
  Polio 3 (OPV3/IPV) | 68.00 | 60.87
  DTP 1 | 100.00 | 95.65
  DTP 2 | 96.00 | 86.96
  DTP 3 | 84.00 | 69.57
  PCV 1 | 92.00 | 86.96
  PCV 2 | 88.00 | 78.26
  PCV 3 | 84.00 | 60.87
  RTR 1 | 76.00 | 78.00
  RTR 2 | 72.00 | 69.57

4. Secondary Outcome: Median Number of Days Children Remain Unvaccinated for Each Vaccine in Intervention Versus Control Arm
Time Frame: Follow-up (up to 6 months post-birth; up to 9 months post-baseline)
Population: Data not collected on 13 participants.
Measure: Median (Full Range); unit: days
Arm/Group | Pregnant Women Receiving VISTA Counseling | Pregnant Women Receiving Usual Care
Number analyzed (Participants) | 25 | 23
days
  BCG | 6.5 [0 to 32] | 12 [2 to 46]
  Polio 0 | 6 [0 to 12] | 8.5 [0 to 33]
  Polio 1 | 5 [-3 to 141] | 3 [-2 to 31]
  Polio 2 | 8 [1 to 78] | 13 [4 to 40]
  Polio 3 | 19 [9 to 51] | 14 [7 to 61]
  Polio IPV | 15 [5 to 59] | 19.5 [4 to 34]
  DTP 1 | 3 [-3 to 24] | 3 [-2 to 31]
  DTP 2 | 9.5 [1 to 59] | 12 [1 to 40]
  DTP 3 | 14.5 [5 to 59] | 17 [4 to 61]
  PCV 1 | 3 [-3 to 24] | 4 [-2 to 31]
  PCV 2 | 9.5 [1 to 59] | 13 [1 to 40]
  PCV 3 | 14.5 [5 to 59] | 17 [4 to 61]
  RTR 1 | 5 [-3 to 41] | 5 [-2 to 58]
  RTR 2 | 20.5 [1 to 59] | 12 [1 to 40]

5. Secondary Outcome: Percentage of Checklist Items Completed During Counseling in VISTA Intervention Arm
Time Frame: Baseline
Population: Outcome measure only applies to the VISTA arm.
Measure: Mean (Full Range); unit: percentage of items
Arm/Group | Pregnant Women Receiving VISTA Counseling | Pregnant Women Receiving Usual Care
Number analyzed (Participants) | 29 | 0
percentage of items | 90.17 [70 to 100] |

6. Secondary Outcome: Mean Number of Minutes Spent Delivering Counseling Per Woman in VISTA Intervention Arm
Time Frame: Baseline
Population: Outcome measure only applies to the VISTA arm.
Measure: Mean (Full Range); unit: minutes
Arm/Group | Pregnant Women Receiving VISTA Counseling | Pregnant Women Receiving Usual Care
Number analyzed (Participants) | 29 | 0
minutes | 15.86 [10 to 24] |

7. Secondary Outcome: Number of Women in the VISTA Intervention Arm Who Say That the Information Provided by the Community Health Worker (CHW) is Helpful
Time Frame: Baseline
Population: Outcome measure only applies to the VISTA arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women Receiving VISTA Counseling | Pregnant Women Receiving Usual Care
Number analyzed (Participants) | 29 | 0
Participants | 28 |

8. Secondary Outcome: Number of Women in the VISTA Intervention Arm Who Say That the Information Provided by the Community Health Worker (CHW) Reduced Their Concerns About Vaccinations
Time Frame: Baseline
Population: Outcome measure only applies to the VISTA arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women Receiving VISTA Counseling | Pregnant Women Receiving Usual Care
Number analyzed (Participants) | 29 | 0
Participants | 24 |

9. Secondary Outcome: Number of Women in the VISTA Intervention Arm Who Say That the Community Health Worker (CHW) Helped Them Understand Why Children Needed Vaccines
Time Frame: Baseline
Population: Outcome measure only applies to the VISTA arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women Receiving VISTA Counseling | Pregnant Women Receiving Usual Care
Number analyzed (Participants) | 29 | 0
Participants | 26 |

10. Secondary Outcome: Number of Women in the VISTA Intervention Arm Who Say That the Community Health Worker (CHW) Answered Most of Their Questions
Time Frame: Baseline
Population: Data not collected.
Arm/Group | Pregnant Women Receiving VISTA Counseling | Pregnant Women Receiving Usual Care
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Number of Women in the VISTA Intervention Arm Who Say That the Community Health Worker (CHW) Was Respectful
Time Frame: Baseline
Population: Outcome measure only applies to the VISTA arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women Receiving VISTA Counseling | Pregnant Women Receiving Usual Care
Number analyzed (Participants) | 29 | 0
Participants | 28 |

12. Secondary Outcome: Number of Women in the VISTA Intervention Arm Who Say That the Community Health Worker (CHW) Explained Things in Terms They Could Understand
Time Frame: Baseline
Population: Outcome measure only applies to the VISTA arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women Receiving VISTA Counseling | Pregnant Women Receiving Usual Care
Number analyzed (Participants) | 29 | 0
Participants | 27 |

13. Secondary Outcome: Number of Women in the VISTA Intervention Arm Who Were Satisfied With Their Conversation With the Community Health Worker (CHW)
Time Frame: Baseline
Population: Outcome measure only applies to the VISTA arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women Receiving VISTA Counseling | Pregnant Women Receiving Usual Care
Number analyzed (Participants) | 29 | 0
Participants | 28 |

14. Secondary Outcome: Number of Women in the VISTA Intervention Arm Who Say They Are Comfortable Vaccinating Their Child
Time Frame: Baseline
Population: Outcome measure only applies to the VISTA arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women Receiving VISTA Counseling | Pregnant Women Receiving Usual Care
Number analyzed (Participants) | 29 | 0
Participants | 29 |

15. Secondary Outcome: Number of Women in the VISTA Intervention Arm Who Say They Will Speak With the CHW Again
Time Frame: Baseline
Population: Outcome measure only applies to the VISTA arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women Receiving VISTA Counseling | Pregnant Women Receiving Usual Care
Number analyzed (Participants) | 29 | 0
Participants | 28 |

16. Secondary Outcome: Number of Women in the VISTA Intervention Arm Who Say They Would Refer the CHW to Their Friends and Family
Time Frame: Baseline
Population: Outcome measure only applies to the VISTA arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Pregnant Women Receiving VISTA Counseling | Pregnant Women Receiving Usual Care
Number analyzed (Participants) | 29 | 0
Participants | 28 |

ADVERSE EVENTS:
Time Frame: Follow-up (up to 6 months post-birth; up to 9 months post-baseline)
Arm/Group | Pregnant Women Receiving VISTA Counseling | Pregnant Women Receiving Usual Care
All-Cause Mortality (participants affected / at risk) | 0/30 | 1/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
Vaccination data for one child in the usual care group was uninterpretable, hence, excluded from assessment of vaccination timeliness outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-02): https://cdn.clinicaltrials.gov/large-docs/86/NCT04421586/Prot_SAP_000.pdf